CLINICAL TRIAL: NCT02897752
Title: Clinical Effects of Peroneal Nerve Functional Electrical Stimulation (WalkAide[R]) for the Lower Extremities in Chronic Stroke Patients With Hemiplegia: A Multicenter, Prospective, Randomized Controlled Trial
Brief Title: Clinical Effects of Peroneal Nerve Functional Electrical Stimulation (WalkAide[R]) for Chronic Stroke Patients
Acronym: PLEASURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Moji Medical Center, Kyusyu Rosai Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIORTHO1523; UMIN-CTR (Other: UMIN000020458)
Record Dates: First submitted 2016-08-05; First posted 2016-09-13 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Stroke
Keywords: stroke; Rehabilitation; WalkAide (WA); Functional Electrical Stimulation (FES)
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WalkAide (Experimental)
  Interventions: Device: gait training with WA
- Usual gait Training (Active Comparator)
  Interventions: Other: usual gait training

INTERVENTIONS:
Device: gait training with WA — Thirty seven units (1 unit=20 minutes) of gait training with WA by a physical therapist for the WA group for 4 weeks (+/- 1 week). Thirteen and 24 of the 37 units are training by a physical therapist and self-training, respectively.
  Arms: WalkAide
Other: usual gait training — Thirty seven units of usual gait training by a physical therapist for the UT group for 4 weeks (+/- 1 week). Thirteen and 24 of the 37 units are training by a physical therapist and self-training, respectively.
  Arms: Usual gait Training

SUMMARY:
RATIONALE:

The previous study resulted that the gait training using Functional Electrical Stimulation (FES) improved the ankle joint function and the walking ability for the chronic stroke patients with foot drop.

In addition, the further exploratory study in multicenter obtained the result that the training with WA were especially good adaptation to the patients who have slight paralysis and can walk independently.

PURPOSE:

This multicenter prospective trial is studying to reveal whether the gait training with the WalkAide[R](WA) for chronic stroke patients who can walk independently is superior to gait training with a physical therapist.

DETAILED DESCRIPTION:
OBJECTIVE:

To reveal whether gait training with the WA for chronic stroke patients who can walk independently (Functional Ambulation Classification [FAC] 5 or 6) is superior to gait training with a physical therapist.

OUTLINE:

This is a multicenter study. Patients continue gait training with WA or without WA for 4 weeks. The effect of rehabilitation is evaluated by 6 Minute Walk Test without device.

ELIGIBILITY:
Inclusion Criteria:

* 1)First-ever hemiplegic patients 4 months after the stroke onset
* 2)Patients whose the lower extremity paralysis is estimated to be stage IV, V or VI according to the Brunnstrom stage
* 3)Patients whose spasticity of the plantar flexor muscle is estimated at 2 or less according to the Modified Ashworth Scale
* 4)Patients whose ankle dorsiflexion range of motion is 0 degree or more
* 5)Patients whose gait performance is estimated to be 5 or 6 according to the FAC
* 6)Patients who can understand the purpose and instructions of this study and complete the training
* 7)Patients who agree to participate in this study and provide their written informed consent

Exclusion Criteria:

* 1)Patients whose ankle dorsiflexion is not induced by the WA due to peripheral neuropathy
* 2)Patients who are contraindicated for the WA (e.g., patients with a metallic implant or implantable medical electrical equipment such as a cardiac pacemaker, and patients with a previous or suspected history of seizure)
* 3)Patients who underwent Botox treatment in the lower extremities within 3 months of this study registry
* 4)Patients who have nervous system (excluding stroke), cardio-respiratory system, or musculoskeletal system disorders, which may affect gait and training
* 5)Patients who had fallen down within a week prior to the registry and are regarded to be at a high risk of falling down by an attending physician
* 6)Patients whose impairment severities changed between the prior and initial assessments

  * Definition of an alteration

    1. Brunnstrom stage for the lower extremity: Confirm whether the stages of the prior and initial assessments are the same value. If these stages are different, this is considered to be an alteration, and the patient with this alteration should be excluded from the study.
    2. Lower extremity subscale of the Fugl-Meyer Assessment: Confirm whether the change in the score between the prior and initial assessments is 5 or less. If the change is 6 or more, then this is considered to be an alteration, and the patient with this alteration should be excluded from the study.
    3. Functional Ambulation Classification: Confirm whether the categories of the prior and initial assessments are the same value. If these categories are different, then this is considered to be an alteration, and the patient with this alteration should be excluded from the study.
* 7) Patients who are regarded to be ineligible for this study by the principal investigator or co-investigators

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-03-23 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test (6MWT; walking distance during a 6-minute walk with maximum effort) | 4weeks
  An evaluation of the effectiveness of WA-assisted gait training using the 6MWT without any device before and after each intervention in the WA-assisted training group (WA group) and usual training group (UT group).

SECONDARY OUTCOMES:
Lower extremity subscale of the Fugl-Meyer Assessment | 4weeks
  An evaluation of the severity of lower extremity using the total score of lower extremity subscale of the Fugl-Meyer Assessment (perfect score: 34 points).
Muscle strength of the ankle dorsiflexor muscle | 4weeks
  An evaluation of the value(Newton/kg) using the ankle back flexor force of three times measured on average, divided by the weight value.
Ankle dorsiflexion range of motion | 4weeks
  An evaluation of range of motion (ROM) as the angle of the ankle succumbed back from the knee joint flexed position in the chair seat position (5 ° increments).
Modified Ashworth Scale for the plantar flexor muscle | 4weeks
  An evaluation of Modified Ashworth Scale (MAS) as the degree of muscle tone six levels ( 0 , 1 , 1+ , 2 , 3 , 4 ) .
  The extent of MAS number indicating the muscle tone degree.
10 Meter Walk Test (10MWT; speed while walking a set distance of 10 m at the patient's preferred speed). | 4weeks
  An evaluation of the effectiveness of WA-assisted gait training using the 10MWT without any device before and after each intervention in the WA and UT groups.
Stroke Impact Scale | 4weeks
  An evaluation of summation score of the total score and physical domain (sixth domain) score.
Adverse event assessment | 4weeks
  A frequency counting of the adverse events. LLT code will be assigned to the reported adverse event using the MedDRA dictionary.
  The origin date of the term until adverse events define the start date of the protocol treatment.

OTHER OUTCOMES:
Improvement of QOL | 4weeks
  Exploratory outcome for improvement of QOL

CONTACTS AND LOCATIONS:
Overall Officials: Kenji Hachisuka, MD, Ph.D, Study Chair — Moji Medical Center, Kyusyu Rosai Hospital, Japan Labour Health Welfare Organization
Locations (24):
- Japan (24):
  - Fukuoka Mirai Hospital, Fukuoka, Fukuoka
  - Nagao Hospital, Fukuoka, Fukuoka
  - Hakujuji Hospital, Fukuoka, Fukuoka
  - Kitakyushu Abeyamakouen Hospital, Kitakyushu, Fukuoka
  - Moji Medical Center, Kyusyu Rosai Hospital, Japan Labour Health Welfare Organization, Kitakyushu, Fukuoka
  - Tobata Rehabilitation Hospital, Kitakyushu, Fukuoka
  - Kitakyushu Yahata Higashi Hospital, Kitakyushu, Fukuoka
  - Shin-Oji Hospital, Kitakyushu, Fukuoka
  - Tochiku Hospital, Kitakyushu, Fukuoka
  - Hospital of the University of Occupational and Environmental Health, Japan, Kitakyushu, Fukuoka
  - Yoshino Hospital, Kitakyushu, Fukuoka
  - Sapporo Shiroishi Memorial Hospital, Sapporo, Hokkaido-prefecture
  - Tokeidai Memorial Hospital, Sapporo, Hokkaido-prefecture
  - Hyogo Prefectural Rehabilitation Central Hospital, Kobe, Hyōgo
  - Yoshida Hospital, Cerebrovascular Research Institute, Kobe, Hyōgo
  - Yamaga Onsen Rehabilitation Hospital, Yamaga, Kumamoto
  - Nichinan Municipal Chubu Hospital, Nichinan, Miyazaki
  - Nagasakikita Hospital, Nishisonogi-gun, Nagasaki
  - Beppu Rehabilitation Center, Beppu, Oita Prefecture
  - Ginowan Memorial Hospital, Ginowan, Okinawa
  - Chuzan Hospital, Okinawa, Okinawa
  - Nanbu-Tokushukai Hospital, Shimajiri-gun, Okinawa
  - Saitama Misato Sogo Rehabilitation Hospital, Misato, Saitama, Saitama
  - Showa Hospital, Shimonoseki, Yamaguchi